CLINICAL TRIAL: NCT02757443
Title: Myocardial Protection With Phosphocreatine in High-RIsk Cardiac SurgEry Patients: a Single-center Randomised Double-blind Placebo-controlled Exploratory Pilot Clinical Trial
Brief Title: Myocardial Protection With Phosphocreatine in High-RIsk Cardiac SurgEry Patients
Acronym: PRISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Principal Investigator, Vladimir Lomivorotov, MD, PhD, Meshalkin Research Institute of Pathology of Circulation
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCr-in-CS
Record Dates: First submitted 2016-04-13; First posted 2016-05-02 (Estimated); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Cardiac Surgical Procedures; Heart Valve Prosthesis Implantation
Keywords: Phosphocreatine; Creatine Phosphate; Neoton; Phosphate, Creatine; Phosphorylcreatine
MeSH Terms: interventions — Phosphocreatine; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phosphocreatine (Experimental): Participants randomly assigned to the phosphocreatine arm receive:
  * after anaesthesia induction 2 g of Phosphocreatine (PCr) prepared in 50 mL of glucose 5% during 30 min intravenous (IV);
  * together with cardioplegia 2.5 g of PCr prepared in 50 mL of glucose 5% and added to every 1 L of cardioplegic solution (Custodiol, Dr. F. KOHLER CHEMIE, GmbH, Germany; concentration = 10 mmol/L);
  * immediately after heart recovery (spontaneous or paced myocardium contraction) after aorta declamping 2 g of PCr prepared in 50 mL of glucose 5% during 30 min IV;
  * immediately after ICU admission 4 g of PCr in 100 mL of glucose 5% during 60 min IV
  Interventions: Drug: Phosphocreatine sodium tetrahydrate after anaesthesia induction; Drug: Phosphocreatine sodium tetrahydrate added to cardioplegia; Drug: Phosphocreatine sodium tetrahydrate after heart recovery; Drug: Phosphocreatine sodium tetrahydrate after ICU admission
- Control (Placebo Comparator): Participants randomly assigned to the placebo arm receive:
  * after anaesthesia induction 50 mL of glucose 5% IV delivered by an identical infusion pump during 30 minutes;
  * together with cardioplegia 50 mL of glucose 5% is added in every 1 L of cardioplegic solution (Custodiol, Dr. F. KOHLER CHEMIE, GmbH, Germany);
  * immediately after heart recovery (spontaneous or paced myocardium contraction) after aorta declamping 50 mL of glucose 5% IV delivered by an identical infusion pump during 30 minutes;
  * immediately after ICU admission 100 mL of glucose 5% IV delivered by an identical infusion pump during 60 minutes
  Interventions: Drug: 5% Glucose after anaesthesia induction; Drug: 5% Glucose; Drug: 5% Glucose after heart recovery; Drug: 5% Glucose after ICU admission

INTERVENTIONS:
Drug: Phosphocreatine sodium tetrahydrate after anaesthesia induction — after anaesthesia induction 2 g of Phosphocreatine (PCr) prepared in 50 mL of glucose 5% during 30 min intravenous (IV)
  Other Names: Neoton
  Arms: Phosphocreatine
Drug: 5% Glucose after anaesthesia induction — after anaesthesia induction 50 mL of glucose 5% IV delivered by an identical infusion pump during 30 minutes
  Other Names: Dextrose
  Arms: Control
Drug: Phosphocreatine sodium tetrahydrate added to cardioplegia — together with cardioplegia 2.5 g of PCr prepared in 50 mL of glucose 5% and added to every 1 L of cardioplegic solution (Custodiol, Dr. F. KOHLER CHEMIE, GmbH, Germany; concentration = 10 mmol/L)
  Other Names: Neoton
  Arms: Phosphocreatine
Drug: 5% Glucose — together with cardioplegia 50 mL of glucose 5% is added in every 1 L of cardioplegic solution (Custodiol, Dr. F. KOHLER CHEMIE, GmbH, Germany)
  Other Names: Dextrose added to cardioplegia
  Arms: Control
Drug: Phosphocreatine sodium tetrahydrate after heart recovery — immediately after heart recovery (spontaneous or paced myocardium contraction) after aorta declamping 2 g of PCr prepared in 50 mL of glucose 5% during 30 min IV
  Other Names: Neoton
  Arms: Phosphocreatine
Drug: 5% Glucose after heart recovery — immediately after heart recovery (spontaneous or paced myocardium contraction) after aorta declamping 50 mL of glucose 5% IV delivered by an identical infusion pump during 30 minutes
  Other Names: Dextrose
  Arms: Control
Drug: Phosphocreatine sodium tetrahydrate after ICU admission — immediately after ICU admission 4 g of PCr in 100 mL of glucose 5% during 60 min IV
  Other Names: Neoton
  Arms: Phosphocreatine
Drug: 5% Glucose after ICU admission — immediately after ICU admission 100 mL of glucose 5% IV delivered by an identical infusion pump during 60 minutes
  Other Names: Dextrose
  Arms: Control

SUMMARY:
There is evidence on the role of the phosphotransfer system in the energy metabolism of the heart, with altered energetics playing an important role in the mechanisms of heart failure. Phosphocreatine plays an important part in the energy heart system. The investigators have just performed a systematic review and meta-analysis of randomized controlled trials (RCTs) and matched studies that compared phosphocreatine with placebo or standard treatment in patients with coronary artery disease or chronic heart failure or in those undergoing cardiac surgery. Patients receiving phosphocreatine had lower all-cause mortality as well as improved cardiac outcomes when compared to the control group, however, the quality of the included studies was low. Thus, the investigators plan to conduct an exploratory high quality RCT to investigate whether providing phosphocreatine compared to placebo improves the myocardial protection in high-risk patients scheduled for cardiac surgery and to determine the best research endpoint for future trials.

ELIGIBILITY:
Inclusion Criteria:

* Double/triple valve lesion that required cardiac surgery with CPB
* Aged 18 years or older
* Signed informed consent

Exclusion Criteria:

* Emergency surgery
* Concomitant coronary artery bypass grafting surgery (CABG) or procedure on any part of the aorta
* Chronic kidney disease of G3-G4-G5 categories according to Kidney Disease: Improving Global Outcomes (KDIGO) criteria (at least one of the following present for > 3 months: glomerular filtration rate ≤ 60 ml/min/1.73 m2, history of kidney transplantation) or solitary kidney (by any reason)
* Known allergy to PCr
* Pregnancy
* Current enrollment into another RCT (in the last 30 days)
* Previous enrollment and randomisation into the PRISE trial
* Administration of PCr in the previous 30 day
* Concomitant radiofrequency/cryo- ablation procedure
* Structural abnormalities or genetic trait point to kidney disease including glomerulonephritis and gout.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Peak concentration of Troponin I | From the randomization to the postoperative day 3 (POD 3)

SECONDARY OUTCOMES:
The need for (yes/no), and dosage (inotropic score) of, inotropic agents | through study completion, an average of 4 weeks
The need for (yes/no), the number of and the dosage of, defibrillation | through study completion, an average of 4 weeks
The incidence of new-onset moderate and severe arrhythmias or cardiac arrest | through study completion, an average of 4 weeks
Cardiac index | at 6 h after ICU admission, and at the beginning of POD 1
Left ventricular ejection fraction | At the beginning of POD 1
Peak serum creatinine concentration | through study completion, an average of 4 weeks
The incidence of acute kidney injury | through study completion, an average of 4 weeks
Sequential Organ Failure Assessment score | through study completion, an average of 4 weeks
Duration of mechanical ventilation | through study completion, an average of 4 weeks
Duration of ICU stay | through study completion, an average of 4 weeks
Duration of hospital stay | through study completion, an average of 4 weeks
30-day all-cause mortality | 30 days after randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny V. Fominskiy, MD PhD, Principal Investigator — Academician EN Meshalkin Novosibirsk Research Institute of Circulation Pathology
Locations (1):
- Evgeny Fominskiy, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Horjus DL, Oudman I, van Montfrans GA, Brewster LM. Creatine and creatine analogues in hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2011 Nov 9;2011(11):CD005184. doi: 10.1002/14651858.CD005184.pub2. PMID 22071819
- [Background] Strumia E, Pelliccia F, D'Ambrosio G. Creatine phosphate: pharmacological and clinical perspectives. Adv Ther. 2012 Feb;29(2):99-123. doi: 10.1007/s12325-011-0091-4. PMID 22297802
- [Background] Landoni G, Zangrillo A, Lomivorotov VV, Likhvantsev V, Ma J, De Simone F, Fominskiy E. Cardiac protection with phosphocreatine: a meta-analysis. Interact Cardiovasc Thorac Surg. 2016 Oct;23(4):637-46. doi: 10.1093/icvts/ivw171. Epub 2016 Jun 17. PMID 27318357
- [Derived] Lomivorotov V, Merekin D, Fominskiy E, Ponomarev D, Bogachev-Prokophiev A, Zalesov A, Cherniavsky A, Shilova A, Guvakov D, Lomivorotova L, Lembo R, Landoni G. Myocardial protection with phosphocreatine in high-risk cardiac surgery patients: a randomized trial. BMC Anesthesiol. 2023 Nov 29;23(1):389. doi: 10.1186/s12871-023-02341-4. PMID 38030971